CLINICAL TRIAL: NCT06159231
Title: Fractional Flow Reserve-guided Percutaneous Coronary Intervention Plus Optimal Medical Treatment Versus Optimal Medical Treatment Alone in Patients with Stable Coronary Artery Disease - FAME II, a 10-year Follow-up Study.
Brief Title: FAME II-10-year Follow-Up
Acronym: FAME2-10yFU
Status: Completed | Type: Observational
Sponsor: CoreAalst BV (Industry)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: CRI-086
Record Dates: First submitted 2023-03-30; First posted 2023-12-06 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The FAME-II trial was a prospective, multicenter, multinational, multi-continental, randomized clinical trial with an 'all comers' design.

The overall purpose of the FAME-II trial was to compare the clinical outcomes, safety and cost-effectiveness of FFR-guided PCI plus optimal medical treatment (OMT) versus OMT alone in patients with stable coronary artery disease and in whom both PCI and medical treatment can be considered on the basis of the presently existing scientific evidence.

FAME-II was conducted from 2009 to 2012 and 1-year, 2-year and 5-year results have been published.

The purpose of this 10-Year Follow-up is to evaluate the 10-year major adverse cardiac event rate (MACE, defined as all-cause death, documented myocardial infarction, unplanned hospitalization leading to urgent revascularization).

Patients will have to sign a specific informed consent for the present 10-year follow-up.

This study will be conducted for about approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with

   1. stable angina pectoris (Canadian Cardiovascular Society Class [CCS] 1, 2, 3)
   2. or, angina pectoris CCS class 4 subsequently stabilized medically (minimum 7 days) or,
   3. atypical chest pain or no chest pain but with documented silent ischemia on non-invasive testing.
2. In whom at least one stenosis was present of at least 50% in one major native epicardial coronary artery with a diameter of at least 2.5 mm and supplying viable myocardium
3. Eligible for PCI
4. Signed written informed consent was obtained. Patients will have to sign a specific informed consent for the present 10-year follow-up.

Exclusion Criteria:

1. Patients in whom the preferred treatment is CABG
2. Patients with left main coronary artery disease requiring revascularization
3. Patients with a recent (less than 1 WEEK) STEMI or Non-STEMI
4. Prior CABG
5. Contra-indication to dual antiplatelet therapy
6. LVEF < 30%
7. Severe LV hypertrophy (defined as a septal wall thickness at echocardiography of more than 13 mm)
8. Planned need for concomitant cardiac surgery (e.g., valve surgery or resection of aortic or left ventricular aneurysm etc.)
9. Extremely tortuous or calcified coronary arteries precluding FFR measurements
10. A life expectancy of less than 2 years
11. Age under 21
12. Pregnancy or intention to become pregnant during the course of the trial
13. Refusal or inability to sign an informed consent. Mental condition (psychiatric or organ cerebral disease) rendering the subject unable to understand the nature, scope, and possible consequences of the trial or mental retardation or language barrier such that the patient is unable to give informed consent
14. Potential for non-compliance towards the requirements in the trial protocol (especially the medical treatment) or follow-up visits
15. Participation or planned participation in another cardiovascular clinical trial before two year follow-up is completed

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that were enrolled in the original FAME2 study, i.e. consecutive patients with stable clinical condition and angiographically defined one-, two, or three-vessel coronary artery disease and amenable for PCI
Sampling Method: Non-Probability Sample
Enrollment: 888 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
The rate of major adverse cardiac events after 10 years of follow-up | 10 years
  10-year major adverse cardiac event rate (MACE, defined as all-cause death, documented myocardial infarction, unplanned hospitalization leading to urgent revascularization).

SECONDARY OUTCOMES:
Comparison of the rate of all-cause death between randomization arms (of the original FAME2 study). | 10 years
  Comparison of the rate of all-cause death between randomization arms (of the original FAME2 study).
Comparison of the rate of documented myocardial infarction between randomization arms (of the original FAME2 study). | 10 years
  Comparison of the rate of documented myocardial infarction between randomization arms (of the original FAME2 study).
Comparison of the rate of unplanned hospitalization leading to urgent revascularization between randomization arms (of the original FAME2 study). | 10 years
  Comparison of the rate of unplanned hospitalization leading to urgent revascularization between randomization arms (of the original FAME2 study).

CONTACTS AND LOCATIONS:
Locations (16):
- United States (3):
  - Stanford University Medical Center, Stanford, California
  - Atlanta VA Medical Center, Decatur, Georgia
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
- Cardiovascular Center Aalst, Aalst, Belgium
- Czechia (2):
  - Masaryk University - Dept. of Internal Cardiology Medicine, Brno, Moravia
  - Nemocnice Na Homolce, Prague
- Rigshospitalet, Copenhagen, Denmark
- Hopital Cardiovasculaire et Pneumologique Louis Pradel, Bron, Lyon, France
- Germany (2):
  - Universität Leipzig Herzzentrum, Leipzig, Saxony
  - München Klinikum Innenstadt, München
- Gottsegen Hungarian Institute of Cardiology, Budapest, Budapest, Hungary
- Azienda Ospedaliera Universitaria S. Anna (Ferrara), Cona, Ferrara, Italy
- Catharina Ziekenhuis, Eindhoven, North Brabant, Netherlands
- Clinical Hospital Center Kragujevac, Kragujevac, Šumadija, Serbia
- Sweden (2):
  - Sodersjukhuset, Stockholm, Stockholm County
  - Universitestssjukhuset i Örebro, Örebro, Örebro County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Collet C, Mahendiran T, Fearon WF, Mizukami T, Munhoz D, Pijls NHJ, Tonino PAL, Barbato E, Piroth Z, Sreckovic M, Thiele H, El Farissi M, Witt N, Rioufol G, Kala P, Engstrom T, Mavromatis K, Frobert O, Verlee P, Brunner S, Mates M, Jagic N, Campo G, Pardaens S, Ikeda K, Pereira TV, da Costa BR, Fournier S, De Bruyne B, Juni P. Fractional flow reserve-guided percutaneous coronary intervention versus medical therapy for stable coronary artery disease: long-term results of the FAME 2 trial. Nat Med. 2026 Jan 15. doi: 10.1038/s41591-025-04132-5. Online ahead of print. PMID 41540107